CLINICAL TRIAL: NCT06629662
Title: Robotic Versus Laparoscopic Sleeve Gastrectomy: Prospective Randomized Study.
Brief Title: Robotic Versus Laparoscopic Sleeve Gastrectomy
Acronym: SLEEVEROBOP
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Naples (Other)
Responsible Party: Principal Investigator, Antonio Vitiello, MD PhD Researcher, University of Naples
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 187/2023
Record Dates: First submitted 2024-10-03; First posted 2024-10-08 (Actual); Last update posted 2025-04-03 (Actual); Status verified 2024-10

CONDITIONS: Robotic Surgery
Keywords: Robotic surgery; Sleeve Gastrectomy; Bariatric surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Laparoscopic sleeve gastrectomy (Active Comparator): Patients undergoing traditional sleeve gastrectomy
  Interventions: Procedure: Sleeve gastrectomy
- Robotic sleeve gastrectomy (Active Comparator): Sleeve gastrectomy with DaVinci robot
  Interventions: Procedure: Sleeve gastrectomy

INTERVENTIONS:
Procedure: Sleeve gastrectomy — Sleeve gastrectomy with laparoscopic or robotic approach

SUMMARY:
Sleeve gastrectomy is the most commonly performed bariatric procedures. Robotic surgery seems to add more precision to the surgical interventions. However, robotic bariatric procedures appear to be burdened by longer operative time.

Aim of the investigators is to prospectively and randomly submit patients suffering from obesity to robotic or laparoscopic surgery in order to compare outcomes.

ELIGIBILITY:
Inclusion Criteria:

* According to IFSO (International Federation for the Surgery of Obesity)/ASMBS (American Society for Metabolic and Bariatric Surgery) 2023 guidelines

Exclusion Criteria:

* Previous bariatric or abdominal surgery

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-11-01 (Estimated)

PRIMARY OUTCOMES:
Operative time | From the Veress needle insertion at the beginning of the surgical intervention to the last skin stich
  Operative time in minutes (Docking plus console time for the robotic procedures)

SECONDARY OUTCOMES:
Intraoperative bleeding | From the Veress needle insertion at the beginning of the surgical intervention to the last skin stich
  Bleeding during the surgical procedure
Postoperative bleeding | From the end of the procedure to postoperative day 30
  Bleeding after the end of the procedure
Conversion to Laparoscopy | From the Veress needle insertion at the beginning of the surgical intervention to the last skin stich
  Conversion to laparoscopy
Conversion to Laparotomy | From the Veress needle insertion at the beginning of the surgical intervention to the last skin stich
  Conversion to laparotomy
Postoperative Leak | From the end of the procedure to postoperative day 30
  Leak from the staple line
Postoperative Bowel Obstruction | From the end of the procedure to postoperative day 30
  Bowel obstruction
Postoperative nausea | From the end of the procedure to postoperative hour 24
  Postoperative nausea measured with a Visuo Analogic Scale (VAS) from 0 (no nausea) to 10 (not tolerable nausea)
Postoperative vomit | From the end of the procedure to postoperative hour 24
  Postoperative vomit measured with a Visuo Analogic Scale (VAS) from 0 (no nausea) to 10 (not tolerable vomit)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Naples Federico II, Naples, Italy, Italy

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol